CLINICAL TRIAL: NCT00445419
Title: A Phase I Single-blind Randomised Placebo Controlled Dose Escalating Study of One Virosome Formulated CD4 and Two Virosomes Formulated CD8 Hepatitis C Virus (HCV) Vaccine Components (PEV2A and PEV2B) Administered to Healthy Adult Volunteers
Brief Title: Phase I Hepatitis C Vaccine Trial of Virosome-formulated Peptides
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pevion Biotech Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHEPC001; 2006DR1345
Record Dates: First submitted 2007-03-08; First posted 2007-03-09 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2010-02

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C; Liver disease; Viral infection; Virosome; Vaccine; therapeutic vaccine; Chronic hepatitis C virus infection
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Liver Diseases; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: PEV2A PEV2B

SUMMARY:
Pevion Biotech has designed a therapeutic vaccine to treat patients who suffer from chronic hepatitis C virus infection. The vaccine is based on a combination of the PeviPRO and PeviTER platforms using synthetic peptide antigens from the hepatitis C virus. Generally, a cellular immune response by cytotoxic T-lymphocytes (CTL) seems to be crucial in overcoming a hepatitis C virus infection. In-depth research in recent years has shown that the cellular immune response is even more effective when supported by helper T-cells. Pevion Biotech's HCV vaccine candidate utilizes this effect inducing specific CTL responses (PeviTER) together with a supportive helper T cell response (PeviPRO). This virosome-based technological combination in a single product represents a new generation of modular therapeutic vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of both sexes
* Aged between 18 and 45 years
* Free of obvious health problems
* With a BMI between 18.5 and 29.9 are included if they give written informed consent

Exclusion Criteria:

* Chronic or acute illness
* Immunosuppression
* HCV and/or HBV infection
* history of allergic disease
* Pre-existing immune response against peptide of the vaccines

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-12; Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events
Specific cellular immune response by Elispot and FACS

SECONDARY OUTCOMES:
Specific proliferative response
Humoral immunity

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Pantaleo, MD, Principal Investigator — Vaccine and Immunotherapy Center (VIC), Division of Immunology and Allergy, CHUV, Lausanne
Locations (1):
- Vaccine and Immunotherapy Center, CHUV, Lausanne, Switzerland

REFERENCES:
- See also: Click here for more information about this study — http://www.pevion.com